CLINICAL TRIAL: NCT01493427
Title: Multi-Center Study Assessing the Efficacy and Tolerability of TRAVATAN® Solution Without BAK, Containing Polyquad® Preservative (0.004% Travoprost) in Patients Previously on Latanoprost 0.005% or Bimatoprost 0.01% Ophthalmic Solution Monotherapy
Brief Title: Efficacy of Changing to TRAVATAN® From Prior Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RDG-10-298; 2011-000161-13 (EudraCT Number)
Record Dates: First submitted 2011-12-14; First posted 2011-12-16 (Estimated); Results first posted 2014-05-09 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma; OAG; OHT
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TRAVATAN® BAK-free (Experimental): Travoprost 0.004%, 1 drop self-administered to the study eye(s) once daily, every evening at around 8:00 pm, for 12 weeks
  Interventions: Drug: Travoprost 0.004%

INTERVENTIONS:
Drug: Travoprost 0.004% — Travoprost 0.004% without benzalkonium chloride (BAK), containing Polyquad (PQ) preservative
  Other Names: TRAVATAN® BAK-free

SUMMARY:
The purpose of this study was to assess the efficacy and tolerability of TRAVATAN® Solution without benzalkonium chloride (BAK) in patients previously on latanoprost 0.005% or bimatoprost 0.01% ophthalmic solution monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ocular hypertension or open-angle glaucoma in at least one eye.
* Be on either latanoprost 0.005% or bimatoprost 0.01% ophthalmic solution monotherapy (including BAK-containing generics) for at least four weeks prior to Screening visit.
* Would benefit from a switch to TRAVATAN® Solution without BAK containing Polyquad® Preservative due to tolerability issues, in the opinion of the investigator.
* IOP considered to be safe (in the opinion of the investigator), in both eyes, in such a way that assured clinical stability of vision and the optic nerve throughout the study period.
* Willing to discontinue the use of all other ocular hypotensive medications prior to receiving the study medication for the entire course of the study.
* Best corrected Snellen visual acuity of 6/60 (20/200, 1.0 LogMAR) or better in each eye
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known medical history of allergy, hypersensitivity, or poor tolerance to any component of the preparations to be used in this study deemed clinically significant in the opinion of the Principal Investigator.
* Any abnormality preventing reliable applanation tonometry in either eye.
* Severe dry eye or related which has been or currently is being treated with the use of punctal plugs, punctal cautery, Restasis®, or topical ocular corticosteroids.
* Any clinically significant, serious, or severe medical condition.
* Intraocular conventional surgery or laser surgery in either eye less than three months prior to Screening Visit.
* Risk of visual field or visual acuity worsening as a consequence of participation in the study, in the investigator's best judgment.
* Progressive retinal or optic nerve disease from any cause.
* Women who are pregnant, lactating.
* Women not using reliable means of birth control.
* Use of any systemic medication known to affect IOP which has not been on stable course for at least 7 days prior to Screening Visit.
* Any clinically significant, serious, or severe medical condition.
* Participation in any other investigational study within 30 days of Screening Visit.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2011-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Severine Durier, Pharm.D, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 15 investigative sites located in Europe: Belgium (2); Spain (6); Italy (4); Sweden (3).
Pre-assignment Details: Of the 202 subjects enrolled, 1 subject was exited as a screen failure and 2 subjects withdrew consent prior to dosing. This reporting group includes all subjects who instilled at least one dose of the test article (199).
Period: Overall Study
Arm/Group | TRAVATAN® BAK-free
Started | 199
Completed | 179
Not Completed | 20
Not completed — Adverse Event | 10
Not completed — Personal Reasons | 4
Not completed — Lost to Follow-up | 2
Not completed — Inability to Follow Instructions | 2
Not completed — Other | 2

BASELINE CHARACTERISTICS:
Population: This reporting group includes all subjects who instilled at least one dose of the test article
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 82

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Intraocular Pressure (IOP) at 12 Weeks From Prior Therapy (Baseline)
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). A more negative change indicates a greater amount of improvement. One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Baseline, Week 12
Population: The Full Analysis Set (FA) included all subjects who instilled at least one drop of study product and who had primary endpoints measures available for at least one on-therapy study visit (N=187). Here, "n" is the number of participants with non-missing values at the specific time point.
Measure: Mean (Standard Deviation); unit: millimeters mercury (mmHg)
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 187
millimeters mercury (mmHg)
  Baseline | 17.0 (3.3)
  Change from Baseline at Week 12 (n=178) | -1.16 (2.65)

2. Secondary Outcome: Percentage of Patients With Target IOP (≤18 mmHg) at 12 Weeks
Description: IOP (fluid pressure inside the eye) was measured by Goldmann applanation tonometry. A higher IOP can be a greater risk for developing glaucoma or glaucoma progression (leading to optic nerve damage). One eye was chosen as the study eye, and only data from the study eye were used for the efficacy analysis.
Time Frame: Week 12
Population: The Full Analysis Set (FA) included all subjects who instilled at least one drop of study product and who had primary endpoints measures available for at least one on-therapy study visit.
Measure: Number; unit: Percentage of participants
Arm/Group | TRAVATAN® BAK-free
Number analyzed (Participants) | 187
Percentage of participants | 81.2

ADVERSE EVENTS:
Time Frame: Adverse event data were collected and reported in the eCRF at each visit from time of first drug instillation to Week 12. Adverse events were collected for the duration of the study (1 year, 2 months).
Description: This reporting group includes all subjects who instilled at least one dose of the test article.
Arm/Group | TRAVATAN® BAK-free
Serious Adverse Events (participants affected / at risk) | 4/199
Other Adverse Events (participants affected / at risk) | 0/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TRAVATAN® BAK-free (N=199)
Upper gastrointestinal hemmorhage (Gastrointestinal disorders) | 1
Pneumonia pneumococcal (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Cholelithiasis (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.